CLINICAL TRIAL: NCT02590562
Title: A Multi-center Cross-sectional Study on Treatment Patterns and Patient Characteristics in Rheumatoid Arthritis (RA) Patients Treated by Biological DMARDs in China
Brief Title: An Observational Study to Describe in Routine Clinical Practice the Treatment Patterns of Usage of Biological DMARDs in RA Patients.
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28487
Record Dates: First submitted 2015-10-16; First posted 2015-10-29 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- RA patients treated with routine clinical practice: Describe in routine clinical practice the treatment patterns of usage of biological DMARDs in patients suffering from RA including frequency of monotherapy, biological DMARDs usage status (types, dosage), concomitant DMARDs usage information (type and dosage)
  Interventions: Other: Routine clinical practice

INTERVENTIONS:
Other: Routine clinical practice

SUMMARY:
This observational study will describe the treatment patterns of usage of biological DMARDs in routine clinical practice and the demographics and RA disease characteristics in patients suffering from rheumatoid arthritis. Patients will be recruited and examined the same day when recruited. There will be no follow up visit or treatment period only one visit in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Patients with a diagnosis of RA according to the revised ACR criteria.
* Patients receiving treatment of launched biological DMARDs.

Exclusion Criteria:

* Patients who received biological DMARDs due to clinical trials or biologics not launched.
* Patients who are considered not appropriate for study due to other reasons at physicians' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include RA patients (according to ACR criteria) who are experiencing biologic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- China (15):
  - Peking University First Hospital, Beijing
  - Beijing Jishutan Hospital; Rheumatology & Immunology, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - China-Janpan Friendship Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Guanghua Hospital of Integrated Traditional Chinese and Western Medicine ( Guanghua Hospital), Shanghai
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin (天津)
  - Xinjiang Uygur Autonomous Region People Hospital, Ürümqi
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Population: Participants diagnosed with rheumatoid arthritis (RA) according to American College of Rheumatology (ACR) 1987 criteria who were using biological disease-modifying anti-rheumatic drugs (DMARDs) approved in China for RA treatment were observed at the single study visit (enrollment visit).
Period: Overall Study
Arm/Group | Overall Population
Started | 808
Completed | 802
Not Completed | 6
Not completed — Did Not Meet the Inclusion Criteria | 6

BASELINE CHARACTERISTICS:
Population: Overall Population: Participants who met all inclusion criteria, diagnosed with RA according to ACR 1987 criteria and were using biological DMARDs approved in China for RA treatment.
Groups:
- Overall Population: Participants diagnosed with RA according to ACR 1987 criteria who were using biological DMARDs approved in China for RA treatment were observed at the single study visit (enrollment visit).
Arm/Group | Overall Population
Number analyzed (Participants) | 802
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was available for 800 participants only; age was missing for 2 participants who were thus not included in the age results.
  years | 49.0 (13.89)
Age, Customized [Number; unit: participants] — Age was available for 800 participants only; age was missing for 2 participants who were thus not included in the age results.
  participants
    less than or equal to (<=) 20 years | 12
    greater than (>) 20 to <=40 years | 201
    >40 to <=60 years | 402
    >60 years | 185
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 652
  Male | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Biological Agent as Monotherapy or in Combination With Conventional Synthesis Disease-modifying Anti-rheumatic Drugs (csDMARDs) Therapy
Description: Biological agent monotherapy meant participants using a biological agent without concomitant csDMARDs. Biological agent monotherapy included biological agent only, biological agent + glucocorticoid, biological agent + non-steroidal anti-inflammatory drugs [NSAIDs], and biological agent + glucocorticoid + NSAIDs.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 802
participants
  Biological agent only | 44
  Biological agent+ glucocorticoid | 9
  Biological agent + NSAIDs | 26
  Biological agent + glucocorticoid + NSAIDs | 5
  Biological agent concomitant with csDMARDs | 718

2. Primary Outcome: Number of Participants Receiving a Biological Agent Concomitant With Other Drugs
Description: Number of participants receiving treatment of a biological agent concomitant with the following drugs: glucocorticoid, NSAIDs, other external medicine, or concomitant glucocorticoid and concomitant NSAIDs. The same participant could use 2 or 3 of concomitant glucocorticoid, NSAIDs and other external medicine.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 802
participants
  Concomitant with glucocorticoid | 238
  Concomitant with NSAIDs | 450
  Concomitant with glucocorticoid and NSAIDs | 137
  Concomitant other external medicine | 153

3. Primary Outcome: Number of Participants Receiving a Biological Agent as Monotherapy by Types of Biological Agents
Description: Number of participants who received a biological agent as monotherapy is presented by biological agent (adalimumab, tocilizumab, etanercept, and infliximab).
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 84
participants
  Adalimumab | 4
  Tocilizumab | 8
  Etanercept | 63
  Infliximab | 9

4. Primary Outcome: Average Weekly Dose of Treatment for Each Biological Agent
Description: Average weekly dose of treatment of each biological agent (adalimumab, tocilizumab, etanercept, or infliximab) is presented.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure. n = participants with specified treatment of biological agent.
Measure: Mean (Standard Deviation); unit: milligrams (mg) per week
Arm/Group | Overall Population
Number analyzed (Participants) | 783
milligrams (mg) per week
  Adalimumab (n=60) | 20.1 (6.41)
  Tocilizumab (n=136) | 94.5 (21.90)
  Etanercept (n=534) | 38.2 (15.64)
  Infliximab (n=53) | 33.1 (23.55)

5. Primary Outcome: Average Duration of Treatment for Each Biological Agent
Description: Average duration of treatment of each biological agent (adalimumab, tocilizumab, etanercept, or infliximab) is presented.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. n = participants with specified treatment of biological agent.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Overall Population
Number analyzed (Participants) | 802
weeks
  Adalimumab (n=60) | 12.7 (19.39)
  Tocilizumab (n=138) | 4.7 (7.48)
  Etanercept (n=535) | 25.5 (47.02)
  Infliximab (n=69) | 34.5 (39.07)

6. Primary Outcome: Number of Participants With Previous Use of the Same Biological Agent
Description: Participants who used the same biological agent in the past and were using that same biological agent at the time of study enrollment.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 802
participants | 58

7. Primary Outcome: Number of Participants With Reasons for Switching Types of Biological Agent Who Used a Different Biological Agent in the Past
Description: Participants who used a different biological agent in the past and switched are shown by reason for switching. One participant could have switched types of biological agent due to multiple reasons.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 93
participants
  Adverse reaction | 13
  Economic reasons | 10
  Unsatisfactory efficacy | 54
  Improvement of the disease | 10
  Inconvenient administration | 2
  Voluntarily discontinuation | 7
  Other reasons | 6

8. Primary Outcome: Average Weekly Dose of Each Concomitant Glucocorticoid
Description: Average weekly dose of each concomitant glucocorticoid (prednisone acetate, oral; betamethasone [BMZ] dipropionate and betamethasone sodium phosphate, intra-articular (IA) injection; and methylprednisolone, intravenous drip infusion, oral) is presented.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure. n = participants with specified concomitant glucocorticoid treatment.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Overall Population
Number analyzed (Participants) | 235
mg/week
  Prednisone acetate, oral (n=174) | 57.8 (31.93)
  BMZ dipropionate and BMZ sodium phosphate, IA(n=2) | 3.8 (4.54)
  Methylprednisolone, intravenous drip infusion(n=4) | 638.8 (368.61)
  Methylprednisolone, oral (n=55) | 59.7 (151.60)

9. Primary Outcome: Average Duration of Treatment With Each Concomitant External Medicine
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure. n = participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Overall Population
Number analyzed (Participants) | 153
weeks
  Baiyi anti-inflammatory analgesic plaster (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Tibetan medicine (n=1) | 24.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Flurbiprofen (n=2) | 4.5 (4.95)
  Compound Nanxing analgesic plaster (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Indirect moxibustion (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Dogskin paste (n=2) | 5.5 (4.95)
  Dogskin plaster (n=1) | 10.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Analgesic plaster for arthritis (n=4) | 90.5 (83.35)
  Hantongle plaster (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Safflower oil (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Wong To Yick Winter Green Oil (n=1) | 40.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Activating collaterals Liniment (n=1) | 4.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Flavored Shuangbai Powder (n=16) | 16.9 (27.99)
  Capsaicin (n=13) | 5.1 (7.13)
  Kilo-Mile Medicine Oil (n=1) | 4.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Qingpeng ointment (n=5) | 40.8 (39.76)
  Shuangbai powder (n=5) | 3.0 (4.47)
  Diclofenac (n=32) | 7.8 (26.39)
  Tianhe ostealgia plaster (n=1) | 4.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Ketoprofen (n=46) | 2.0 (4.06)
  Xiaotong plaster (n=5) | 83.2 (45.62)
  Anti-inflammatory analgesic ointment (n=1) | 1.1 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Antiphlogistic analgesic ointment (n=1) | 5.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Yunnan Baiyao plaster (n=3) | 59.0 (84.54)
  Chinese patent medicine (n=2) | 2.0 (0.00)
  Indometacin (n=1) | 4.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Musk tiger bone plaster (n=1) | 10.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Musk analgesic spray (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Shexiang Zhuanggu plaster (n=1) | 3.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Missing (n=1) | 1.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.

10. Primary Outcome: Number of Participants Using One, Two, or Three (or More) Concomitant csDMARDs
Description: Number of participants using one concomitant csDMARD, two concomitant csDMARDs (methotrexate + hydroxychloroquine [HCQ], methotrexate + salazosulfapyridine [SASP], methotrexate+ leflunomide, SASP + HCQ, and other combinations), or three (or more) concomitant csDMARDs (methotrexate + SASP + HCQ, and other combinations) are presented.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 718
participants
  One csDMARDs | 354
  Two csDMARDs: Methotrexate + HCQ | 129
  Two csDMARDs: Methotrexate + SASP | 7
  Two csDMARDs: Methotrexate+ leflunomide | 83
  Two csDMARDs: SASP + HCQ | 9
  Two csDMARDs: Other combinations | 68
  Three(or more) csDMARDs: Methotrexate + SASP + HCQ | 10
  Three (or more) csDMARDs: Other combinations | 58

11. Primary Outcome: Average Weekly Dose of Each Concomitant csDMARD
Description: One participant could have received multiple concomitant csDMARDs treatment.
Time Frame: Day 1 (enrollment visit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Overall Population
Number analyzed (Participants) | 718
mg/week
  Iguratimod (n=8) | 46.9 (8.84)
  Cyclophosphamide (n=7) | 26.9 (18.68)
  Ciclosporin (n=2) | 75.0 (35.36)
  Methotrexate (n=473) | 1.4 (0.35)
  Leflunomide (n=298) | 15.4 (5.22)
  Chloroquine phosphate (n=1) | 250.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Azathioprine (n=1) | 50.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Sulfasalazine (n=45) | 1753.3 (693.26)
  Mycophenolate mofetil (n=2) | 625.0 (530.33)
  Minocycline (n=1) | 100.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Penicillamine (n=8) | 343.8 (57.86)
  Thalidomide (n=4) | 75.0 (28.87)
  Hydroxychloroquine (n=300) | 340.3 (96.25)

12. Primary Outcome: Average Duration of Treatment With Each Concomitant csDMARD
Description: One participant could have received multiple concomitant csDMARDs treatment.
Time Frame: Day 1 (enrollment visit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Overall Population
Number analyzed (Participants) | 718
weeks
  Iguratimod (n=6) | 260.8 (121.84)
  Cyclophosphamide (n=7) | 251.1 (230.78)
  Ciclosporin (n=2) | 448.0 (554.37)
  Methotrexate (n=468) | 443.7 (845.76)
  Leflunomide (n=296) | 413.4 (578.53)
  Chloroquine phosphate (n=1) | 95.2 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Azathioprine (n=1) | 0.7 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Sulfasalazine (n=45) | 429.1 (1039.86)
  Mycophenolate mofetil (n=2) | 10.2 (4.45)
  Minocycline (n=1) | 210.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Penicillamine (n=8) | 768.8 (1012.51)
  Thalidomide (n=4) | 234.5 (208.79)
  Hydroxychloroquine (n=298) | 261.3 (409.44)

13. Primary Outcome: Average Daily Dose of Each Currently Concomitant NSAIDs
Description: One participant could have received multiple concomitant NSAIDs treatment.
Time Frame: Day 1 (enrollment visit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Overall Population
Number analyzed (Participants) | 450
mg/day
  Imrecoxib (n=20) | 200.0 (0.00)
  Ibuprofen (n=12) | 550.0 (173.21)
  Aceclofenac (n=7) | 157.1 (53.45)
  Lornoxicam (n=6) | 16.0 (0.00)
  Loxoprofen sodium (n=54) | 143.9 (45.28)
  Meloxicam (n=91) | 12.8 (3.45)
  Nimesulide (n=18) | 186.1 (41.32)
  Celecoxib (n=194) | 306.2 (100.07)
  Diclofenac (n=31) | 130.6 (166.55)
  Etoricoxib (n=26) | 86.5 (32.12)
  Indometacin (n=1) | 75.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.

14. Primary Outcome: Average Daily Dose of Each Previously Concomitant NSAIDs
Description: One participant could have received multiple concomitant NSAIDs treatment.
Time Frame: Day 1 (enrollment visit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Overall Population
Number analyzed (Participants) | 98
mg/day
  Ibuprofen (n=8) | 525.0 (148.80)
  Aceclofenac (n=2) | 150.0 (70.71)
  Loxoprofen sodium (n=16) | 135.0 (46.48)
  Meloxicam (n=18) | 13.1 (3.69)
  Nimesulide (n=1) | 200.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.
  Celecoxib (n=39) | 266.7 (95.51)
  Diclofenac (n=12) | 83.3 (40.36)
  Etoricoxib (n=3) | 60.0 (0.00)
  Indometacin (n=1) | 75.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this category.

15. Secondary Outcome: Number Participants With Past Medical History of Concurrent Chronic Disease, Tuberculosis, Hepatitis, and Imaging Manifestations of Joint Damage
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 802
participants
  Concurrent chronic disease | 275
  Tuberculosis history | 2
  Hepatitis history | 8
  Imaging of joint damage | 279

16. Secondary Outcome: Weight
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Overall Population
Number analyzed (Participants) | 799
kilograms | 58.9 (10.55)

17. Secondary Outcome: Height
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Overall Population
Number analyzed (Participants) | 797
centimeters (cm) | 161.6 (6.56)

18. Secondary Outcome: Number of RA Related Operations
Description: RA related operations also included prosthesis.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: RA related operations
Arm/Group | Overall Population
Number analyzed (Participants) | 801
RA related operations | 0.1 (0.34)

19. Secondary Outcome: RA Duration Since Diagnosis
Description: RA duration = (the date of participants signing the informed consent form - date of RA diagnosis + 1) /365.25
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Overall Population
Number analyzed (Participants) | 357
years | 3.2 (5.80)

20. Secondary Outcome: Number of Participants With RA Duration
Description: Number of participants with RA duration of <= 6 months, >6 months and <= 3 years, >3 years and <= 10 years, and 10 years.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 357
participants
  <=6 months | 176
  >6 months and <=3 years | 80
  >3 years and <=10 years | 59
  10 years | 42

21. Secondary Outcome: Number of Participants With Concurrent RA Extra-articular Symptoms
Description: Number of participants with concurrent RA extra-articular symptoms including RA subcutaneous nodule, RA vasculitis, interstitial pneumonia, Felty's syndrome, and other symptoms were presented. One participant could have more than one concurrent RA extra-articular symptoms.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 41
participants
  RA nodule | 18
  Vasculitis | 0
  Interstitial pneumonia | 22
  Felty's syndrome | 0
  Other symptoms | 2

22. Secondary Outcome: Number of Participants With Concurrent Interstitial Lung Disease Using Methotrexate
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 22
participants | 5

23. Secondary Outcome: C-Reactive Protein (CRP) Values
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Overall Population
Number analyzed (Participants) | 344
mg/L | 27.7 (33.91)

24. Secondary Outcome: Number of Participants With Abnormal CRP Values
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Central lab was not used in this study; the definitions of abnormal CRP followed participating hospitals' standardized criteria. Case report form (CRF) collected data as directly "normal" or "abnormal".
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 344
participants | 209

25. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Values
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. A higher rate is consistent with inflammation.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Overall Population
Number analyzed (Participants) | 394
mm/hr | 42.4 (31.10)

26. Secondary Outcome: Number of Participants With Abnormal ESR Values
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. A higher rate is consistent with inflammation. Central lab was not used in this study; the definitions of abnormal ESR followed participating hospitals' standardized criteria. CRF collected data as directly "normal" or "abnormal".
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 394
participants | 276

27. Secondary Outcome: Hemoglobin Values
Description: Hemoglobin levels were measured in gram per liter (g/L). Anemia was defined as an adult male with hemoglobin value <120 g/L or an adult female with hemoglobin value <110 g/L.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Overall Population
Number analyzed (Participants) | 411
g/L | 117.1 (18.78)

28. Secondary Outcome: Number of Participants With Anemia
Description: Anemia was defined as an adult male with hemoglobin value <120 g/L or an adult female with hemoglobin value <110 g/L.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 411
participants | 147

29. Secondary Outcome: Number of Participants With Positive Anti-cyclic Citrullinated Peptide (ACCP) Antibody
Description: ACCP antibodies are important markers of bone erosion in RA. Central lab was not used in this study; the definitions of positive ACCP followed participating hospitals' standardized criteria. CRF collected data as "positive" or "negative" directly.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 173
participants | 144

30. Secondary Outcome: Number of Participants With Positive Rheumatoid Factor (RF)
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. Central lab was not used in this study; the definitions of positive RF followed participating hospitals' standardized criteria. CRF collected data as "positive" or "negative" directly.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 237
participants | 184

31. Secondary Outcome: Triglyceride Values
Description: Normal range for triglyceride is <1.7 millimoles per liter (mmol/L).
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Overall Population
Number analyzed (Participants) | 226
mmol/L | 1.3 (0.71)

32. Secondary Outcome: Number of Participants With Abnormal Triglyceride Values
Description: Normal range for triglyceride is <1.7 mmol/L.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 226
participants | 47

33. Secondary Outcome: Total Cholesterol Values
Description: Normal range for total cholesterol is <5.2 mmol/L.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Overall Population
Number analyzed (Participants) | 233
mmol/L | 4.3 (1.23)

34. Secondary Outcome: Number of Participants With Abnormal Total Cholesterol Values
Description: Normal range for total cholesterol is <5.2 mmol/L.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 233
participants | 35

35. Secondary Outcome: Swollen Joint Count (SJC)
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Overall Population
Number analyzed (Participants) | 802
swollen joint count | 4.8 (6.06)

36. Secondary Outcome: Tender Joint Count (TJC)
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Overall Population
Number analyzed (Participants) | 802
tender joint count | 6.7 (7.21)

37. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) or CRP (mg/dL), and Patient's Global Assessment (PtGA) of disease activity (measured on a 0 to 100 mm Visual Analogue Scale [VAS] where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PtGA of disease activity; DAS28-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(10*CRP+1) + 0.014*PtGA of disease activity. DAS28-ESR was adopted to calculate DAS28 if effective ESR data was available; otherwise DAS28-CRP was adopted to calculate DAS28. Total score range: 0-10, higher score=more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 412
units on a scale | 4.4 (1.52)

38. Secondary Outcome: Number of Participants Experiencing High Disease Activity to Clinical Remission Using the DAS28
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) or CRP (mg/dL), and PtGA of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014*PtGA of disease activity; DAS28-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(10*CRP+1) + 0.014*PtGA of disease activity. DAS28-ESR was adopted to calculate DAS28 if effective ESR data was available; otherwise DAS28-CRP was adopted to calculate DAS28. Total score range: 0-10, higher score=more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 412
participants
  High disease activity | 135
  Moderate disease activity | 174
  Low disease activity | 51
  Remission | 52

39. Secondary Outcome: Clinical Disease Activity Index (CDAI) Scores
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and Physician's Global Assessment (PGA) assessed on 0-10 centimeter (cm) VAS; 0 = no disease activity and 10 = worst disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 801
units on a scale | 20.2 (15.25)

40. Secondary Outcome: Number of Participants Experiencing High Disease Activity to Clinical Remission Using the CDAI
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 801
participants
  High disease activity | 278
  Moderate disease activity | 273
  Low disease activity | 207
  Remission | 43

41. Secondary Outcome: Simplified Disease Activity Index (SDAI)
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity, and CRP (mg/dL). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 343
units on a scale | 27.2 (18.09)

42. Secondary Outcome: Number of Participants Experiencing High Disease Activity to Clinical Remission Using the SDAI
Description: as for outcome 41
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 343
participants
  High disease activity | 158
  Moderate disease activity | 117
  Low disease activity | 56
  Remission | 12

43. Secondary Outcome: Number of Participants With Duration of Treatment of Biological Agent
Description: Number of participants with duration of treatment of biological agent <3 months, >= 3 to <6 months, >= 6 to <12 months, and >= 12 months.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 802
participants
  <3 months | 503
  >=3 to <6 months | 86
  >=6 to <12 months | 96
  >=12 months | 117

44. Secondary Outcome: DAS28 by Duration of Treatment of Biological Agent
Description: as for outcome 38
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure in respective arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duration of Biological Treatment <3 Months: Participants were divided into groups with different duration of treatment according to the months of using biological agent. This group included participants with duration of biological treatment <3 months.
- Duration of Biological Treatment >=3 to <6 Months: Participants were divided into groups with different duration of treatment according to the months of using biological agent. This group included participants with duration of biological treatment >=3 to <6 months.
- Duration of Biological Treatment >=6 to <12 Months: Participants were divided into groups with different duration of treatment according to the months of using biological agent. This group included participants with duration of biological treatment >=6 to <12 months.
- Duration of Biological Treatment >=12 Months: Participants were divided into groups with different duration of treatment according to the months of using biological agent. This group included participants with duration of biological treatment >=12 months.
Arm/Group | Duration of Biological Treatment <3 Months | Duration of Biological Treatment >=3 to <6 Months | Duration of Biological Treatment >=6 to <12 Months | Duration of Biological Treatment >=12 Months
Number analyzed (Participants) | 312 | 35 | 25 | 40
units on a scale | 4.6 (1.45) | 3.5 (1.44) | 3.9 (1.42) | 3.2 (1.40)
Statistical Analysis 1: Comparison: Duration of Biological Treatment <3 Months vs Duration of Biological Treatment >=3 to <6 Months vs Duration of Biological Treatment >=6 to <12 Months vs Duration of Biological Treatment >=12 Months; Test type: Superiority or Other; p < 0.0001, F test

45. Secondary Outcome: DAS28 by Biological Agent as Monotherapy or Combination With csDMARDs
Description: Biological agent monotherapy meant participants using a biological agent without concomitant csDMARDs. DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) or CRP (mg/dL), and PtGA of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014*PtGA of disease activity; DAS28-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(10*CRP+1) + 0.014*PtGA. DAS28-ESR was adopted to calculate DAS28 if effective ESR data was available; otherwise DAS28-CRP was adopted to calculate DAS28. Total score range: 0-10, higher score=more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biological Agent as Monotherapy: Participants were divided into two groups according to whether using biological agent (namely, biological agent concomitant with csDMARDs treatment group and biological agent without csDMARDs treatment group). This group included participants using biological agent without concomitant csDMARDs.
- Biological Agent as Combination With csDMARDs: Participants were divided into two groups according to whether using biological agent (namely, biological agent concomitant with csDMARDs treatment group and biological agent without csDMARDs treatment group). This group included participants using biological agent with concomitant csDMARDs.
Arm/Group | Biological Agent as Monotherapy | Biological Agent as Combination With csDMARDs
Number analyzed (Participants) | 56 | 356
units on a scale | 4.8 (1.76) | 4.3 (1.47)
Statistical Analysis 1: Comparison: Biological Agent as Monotherapy vs Biological Agent as Combination With csDMARDs; Test type: Superiority or Other; p = 0.0108, F test

46. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Activity
Description: PGA of disease activity was measured on a 0 to 10 centimeter (cm) VAS, with 0 cm = no disease activity and 10 cm = extreme disease activity.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Overall Population
Number analyzed (Participants) | 802
cm | 4.2 (2.23)

47. Secondary Outcome: Patient's Global Assessment (PtGA) of Disease Activity
Description: PtGA of disease activity was measured on a 0 to 10 cm VAS, with 0 cm = very well controlled and 10 cm = very poorly controlled.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Overall Population
Number analyzed (Participants) | 801
cm | 4.4 (2.30)

48. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ consists of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question has 4 response options, ranging from "no difficulty" to "unable to do", corresponding to scores from 0 to 3. HAQ total score = sum of each of the 20 items' scores, with a summary score ranging from 0 to 60, where higher score indicates greater disability.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 800
units on a scale | 11.9 (13.44)

49. Secondary Outcome: Participant's Fatigue Assessment
Description: Participants scored the fatigue on 10 cm VAS from 0 = no fatigue to 10 = very fatigue.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Overall Population
Number analyzed (Participants) | 801
cm | 3.7 (2.51)

50. Secondary Outcome: Participant's Pain Assessment
Description: Participants scored the intensity of pain produced by RA on 10 cm VAS from 0 = no pain to 10 = extreme pain.
Time Frame: Day 1 (enrollment visit)
Population: Overall Population. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Overall Population
Number analyzed (Participants) | 801
cm | 4.2 (2.44)

ADVERSE EVENTS:
Time Frame: Day 1 (enrollment visit)
Description: Overall population
Arm/Group | Overall Population
Serious Adverse Events (participants affected / at risk) | 0/802
Other Adverse Events (participants affected / at risk) | 5/802
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Population (N=802)
Abnormal liver function (Hepatobiliary disorders) | 1
Amyosthenia (Musculoskeletal and connective tissue disorders) | 1
Erythra (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.